CLINICAL TRIAL: NCT05065281
Title: Responding to Elder Abuse in GERiAtric Care Educational Intervention for Healthcare Providers: a Non-randomised Stepped Wedge Trial.
Brief Title: Responding to Elder Abuse in GERiAtric Care: Educational Intervention
Acronym: REAGERA edu
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Östergötland (Other)
Collaborators: Linkoeping University (Other Government); Region Jönköping County (Other Government); Linnaeus University (Other); Kamprad Family Foundation (Unknown); Medical Research Council of Southeast Sweden (Other Government)
Responsible Party: Principal Investigator, Johanna Simmons, Principal Investigator, Region Östergötland
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: RÖ-786
Record Dates: First submitted 2021-09-15; First posted 2021-10-04 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Healthy
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Non-randomized stepped wedge cluster trial (incomplete design)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education (Experimental): Participants that have undergone the educational intervention
  Interventions: Other: Education
- Waitlist (No Intervention): Participants still waiting to cross over to intervention arm

INTERVENTIONS:
Other: Education — Training for health care professionals on how to identify and manage cases of elder abuse among their patients
  Arms: Education

SUMMARY:
The prevalence of elder abuse has been reported between 10-15% in international studies. Elder abuse may include both physical, emotional, sexual and financial abuse as well as neglect and it occurs at the hand of both professionals and family members, including adult children and intimate partners. Elder abuse has been associated with psychological ill-health, disability, increased hospitalization, emergency department use and admission to nursing facilities. Elder abuse is however often unknown to health care providers. Older adults are hesitant to disclose abuse and health care providers are often reluctant to ask questions.

In this study an interactive educational model for health care professionals about elder abuse will be tested. The model consist of theoretical lectures, brief films showing patient encounters, group discussions and forum play, a form of participatory theater. Both group discussions and forum play will be using case scenarios as a cornerstone.

The validated questionnaire REAGERA-P will be used for self-reported measures

DETAILED DESCRIPTION:
Please refer to the uploaded study protocol for a detailed description of the study.

ELIGIBILITY:
Inclusion Criteria:

* Employee at one of the clinics participating in the trial
* Work tasks involves direct patient contact, at least part time
* Participation at the training sessions

Exclusion Criteria:

* Only administrative work and no direct patient contact
* Not participating at the training session

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 554 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Change between baseline and follow up concerning asking questions about abuse, as reported in the questionnaire REAGERA-P | Baseline, 6 month follow up, 12 month follow up
  Self-report measure of asking older patients about abusive experience. Will be measure both as a dichotomous value (have ever asked questions during the last 6 months) as well as a frequency measure where participants report how often they have asked patients questions about abuse during the last 6 months (on a scale from 0 to 10 or more)

SECONDARY OUTCOMES:
Change between baseline and follow up concerning awareness of elder abuse and sense of responsibility for identifying victims, as reported in the questionnaire REAGERA-P | Baseline, Immediate post-intervention (number 2), 6 month follow up, 12 month follow up
  1. Self-reported perceived lack of awareness of elder abuse as a barrier toward identifying victims.
  2. Self reported sense of responsibility for asking questions about abuse (own responsibility, professions' responsibility, health care services responsibility)
Change between baseline and follow up concerning level of awareness of abuse in contact with patients, as reported in the questionnaire REAGERA-P | Baseline, 6 or 12 month follow up (different for different clusters)
  Patient case ("Vignette") with indicators of abuse and participants self-report if they think they would have asked the patient questions about abuse
Change between baseline and follow up concerning perceived ability to ask questions about abuse, as reported in REAGERA-P | Baseline, Immediate post-intervention, 6 month follow up, 12 month follow up
  1. Self-reported self-efficacy for asking questions about elder abuse.
  2. Self-reported cause for concern that asking questions will a) lead to a negative reaction from the patient b) negatively impact the patient-provider relationship
Change between baseline and follow up concerning perceived preparedness to manage cases of elder abuse, as reported in REAGERA-P | Baseline, Immediate post-intervention (number 1and 2), 6 months follow up, 12 months follow up
  1. Self-reported self-efficacy for managing cases of elder abuse.
  2. Self-reported cause for concern of not being able to offer the patient a good follow up.
  3. Self-reported collegial support, i.e., knowing which colleague to ask for help if needed when managing cases of elder abuse.
  4. Self-reported knowledge about proper documentation routines
  5. Self-reported knowledge about judicial concerns
Change between baseline and follow up concerning preparedness at the clinic to care for older adults subjected to abuse, as reported in REAGERA-P | Baseline, 6 months follow up, 12 months follow up
  Self-reported evaluation of:
  1. Routines for managing cases of elder abuse at the clinic
  2. Preparedness at the clinic and in society to care for victims of elder abuse.

OTHER OUTCOMES:
Change between baseline and follow up concerning number of elder abuse victims identified at the clinics included in the study, as reported in the medical records | Baseline, 6 month follow up, 12 month follow up
  Anonymous data from the medical records counting the number of older patients treated at each clinic that have been identified as victims of abuse during the last 6 months
Change between baseline and follow up concerning adequate follow up, as reported in the questionnaire REAGERA-P | Baseline, 6 month follow up, 12 month follow up
  Frequency of respondents reporting that identified cases of elder abuse were given adequate follow up
Change between baseline and follow up concerning self-reported hesitancy for asking questions about elder abuse, as reported in the questionnaire REAGERA-P | Baseline, 6 month follow up, 12 month follow up
  Frequency of respondents reporting that they have suspected cases of elder abuse but refrained from asking questions
Degree of changed practice as reported in the questionnaire REAGERA-P | 6 month follow up
  Frequency of participants self-reporting that they have changed their working practices as a result of the educational intervention

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Simmons, MD, PhD, Principal Investigator — Region Östergötland
Locations (4):
- Sweden (4):
  - Region Jönköpings län, Eksjö
  - Region Jönköpings Län, Jönköping
  - Region Östergötland, Linköping
  - Region Östergötland, Norrköping

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make anonymous participant data that underlie results in publications available. However, we are still waiting on final guidelines from the sponsor concerning sharing data and in the unlikely case that the new guidelines prohibit sharing data it will not be shared.
Time Frame: Data will become available alongside publications.
Access Criteria: Will be made available from the researcher upon reasonable request or made available from a public depository.

REFERENCES:
- [Background] Simmons J, Wenemark M, Ludvigsson M. Development and validation of REAGERA-P, a new questionnaire to evaluate health care provider preparedness to identify and manage elder abuse. BMC Health Serv Res. 2021 May 19;21(1):473. doi: 10.1186/s12913-021-06469-2. PMID 34006271
- [Background] Ludvigsson M, Motamedi A, Westerlind B, Swahnberg K, Simmons J. Responding to Elder Abuse in GERiAtric care (REAGERA) educational intervention for healthcare providers: a non-randomised stepped wedge trial. BMJ Open. 2022 May 4;12(5):e060314. doi: 10.1136/bmjopen-2021-060314. PMID 35508341
- See also: Study Protocol — http://dx.doi.org/10.1136/bmjopen-2021-060314

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-02): https://cdn.clinicaltrials.gov/large-docs/81/NCT05065281/Prot_SAP_002.pdf